CLINICAL TRIAL: NCT02377479
Title: Endocrinology Profile in Patients Undergoing Clomiphene, Letrozole, and Combination Clomiphene and Letrozole Cycles
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Study never started
Sponsor: University Hospitals Cleveland Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 043234
Record Dates: First submitted 2015-02-25; First posted 2015-03-03 (Estimated); Last update posted 2022-05-12 (Actual); Status verified 2022-05

CONDITIONS: Infertility
MeSH Terms: conditions — Infertility | interventions — Clomiphene; Letrozole

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Clomiphene alone (Active Comparator): The patient will take 100mg clomiphene orally from cycle days 3-7
  Interventions: Drug: Clomiphene
- Letrozole alone (Active Comparator): The patient will take 5mg Letrozole orally from cycle days 3-7
  Interventions: Drug: Letrozole
- Combination Clomiphene and Letrozole (Experimental): The patient will take a dose of 5mg Letrozole every night and 100mg clomiphene every day after lunch from cycle days 3-7.
  Interventions: Drug: Clomiphene; Drug: Letrozole

INTERVENTIONS:
Drug: Clomiphene — Taken for controlled ovarian hyperstimulation.
  Other Names: Clomid
  Arms: Clomiphene alone; Combination Clomiphene and Letrozole
Drug: Letrozole — Taken for controlled ovarian hyperstimulation
  Other Names: Femara
  Arms: Combination Clomiphene and Letrozole; Letrozole alone

SUMMARY:
The goal of the study is to measure serial hormonal levels in patients undergoing clomiphene, letrozole, and a combination clomiphene and letrozole cycle. This information may help us to optimize less expensive medications for ovulation induction, reduce the number of treatment cycles to achieve a successful pregnancy, and use a medication regimen that may result in fewer multiple gestation pregnancies.

DETAILED DESCRIPTION:
After the initial physician consultation and investigations have been completed, the treatment options will be reviewed with the patient. If the patient chooses ovulation induction with an oral medication, then she will be offered participation in the study.

If she chooses to participate, the patient will then undergo ovulation induction with either clomiphene, letrozole, or a combination of both medications. The patient will be randomized to the order that each medication regimen will be started. Prior to starting each treatment cycle, a serum beta-hCG (serum beta-hCG < 5IU/L) or urine pregnancy test will be performed to rule out pregnancy.

During one treatment cycle, the patient will take 100mg clomiphene orally from cycle days 3-7. This dose is routinely used for ovulation induction in the investigators clinic. Blood work including an estradiol (E2), FSH, inhibin B and LH will be obtained on cycle days 3, 7, and 9. As these lab tests are routinely performed in the investigators REI laboratory, there will be no additional cost to the patient. A baseline follicle count by ultrasound during each treatment cycle will be measured on cycle day 3, and then again on cycle day 12, 13, or 14, depending on the cycle length until the lead follicle is 18mm or greater. Once at least one follicle has reached this mature size, an Ovidrel trigger (250 mcg hCG subcutaneously) will be administered to initiate ovulation. The patient will have an intrauterine insemination (IUI) 36 hours after Ovidrel injection. These procedures are the current standard of care in the investigators fertility center for patients with unexplained infertility.

Ovulation during each treatment cycle will also be confirmed with a serum progesterone measurement >3 nmol/L on cycle day 20-25. This blood test is not always performed, but is a common way to assess ovulation.

If the patient ovulated, a pregnancy test will be performed approximately 2 weeks later. If pregnancy has not occurred, the next medication would be attempted after the patient has a period.

During the second treatment cycle, the patient will take 5mg Letrozole orally from cycle days 3-7. The remainder of the prior protocol for the clomiphene cycle would then be performed. This medication dose and protocol are also the current standard of care in the investigators fertility center.

During the third treatment cycle, the patient will take a dose of 5mg Letrozole every night and 100mg clomiphene every day after lunch from cycle days 3-7. The remainder of the prior protocol for the clomiphene cycle would then be performed. This combination dose would be the experimental portion of the protocol, as it has been done before, but is not currently standard of care in the investigators fertility center.

If the patient does not ovulate despite giving hCG subcutaneously or the lead follicle never reaches >/= 18mm, that treatment cycle will be abandoned. After the patients next period, she will be started immediately on the next treatment cycle.

If, upon failing to ovulate with any of the medication regimens, a subject declines to continue with the next medication and would prefer to go straight to gonadotropin treatment with or without IVF treatment, the subject will still remain as part of the study and only the US and bloodwork values obtained while still involved in the study will be included.

A subject will have completed the study after one cycle of clomiphene, one cycle of letrozole, and one cycle of combination clomiphene/IUI have been achieved. For patients that do not achieve a pregnancy at the end of the study, they will have the option to undergo other fertility treatments that will be discussed with their primary fertility specialist.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-40 years old
* Body mass index (BMI) > 18 kg/m^2 and < 40kg/m^2
* No contraindications to clomiphene or letrozole
* Ovulatory women
* 1 month without any fertility medication

Exclusion Criteria:

* Patients unable to consent for the study
* Patients with polycystic ovarian syndrome or anovulatory women

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2015-03; Primary Completion 2017-03 (Estimated)

PRIMARY OUTCOMES:
The endocrinology profile (LH, FSH, estradiol, inhibin B) during a letrozole, clomiphene, and combination letrozole and clomiphene cycle | 1 month
  The LH, FSH, estradiol, inhibin B levels will be measured on cycle days 3, 7, and 9.

SECONDARY OUTCOMES:
1. Pregnancy rate | 1 month
Ovulation rate | 1 month
Ongoing pregnancy rate (pregnancy with fetal heartbeat > 12 weeks gestational age) | 12 weeks
Miscarriage rate | 10 weeks
Multiple pregnancy rate (twins and higher order multiples) | 6- 8 weeks
Number of mature follicles (>/= 18mm) | 1 month

CONTACTS AND LOCATIONS:
Locations (1):
- University Hospitals Fertility Center, Beachwood, Ohio, United States